CLINICAL TRIAL: NCT01764347
Title: Accuracy of Targeted Biopsies Using MRI-TRUS Fusion Guidance: Pilot Study on Ex Vivo Radical Prostatectomy Specimens
Brief Title: Magnetic Resonance Imaging-Transrectal Ultrasound Fusion Image-Guided Prostate Biopsy Following Radical Prostatectomy in Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4P-10-6; NCI-2012-03037 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-12-21; First posted 2013-01-09 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (MRI-TRUS fusion image-guided biopsy) (Experimental): Patients undergo robotic radical prostatectomy, followed by 3 MRI-TRUS fusion image-guided prostate biopsies.
  Interventions: Procedure: therapeutic conventional surgery; Procedure: ultrasound-guided prostate biopsy; Procedure: magnetic resonance imaging

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Undergo robotic radical prostatectomy
Procedure: ultrasound-guided prostate biopsy — Undergo MRI-TRUS fusion image-guided prostate biopsy
Procedure: magnetic resonance imaging — Undergo MRI-TRUS fusion image-guided prostate biopsy
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This pilot clinical trial studies magnetic resonance imaging (MRI)-transrectal ultrasound (TRUS) fusion image-guided prostate biopsy following radical prostatectomy in patients with prostate cancer. Diagnostic procedures, such as MRI-TRUS fusion image-guided prostate biopsy may help find and diagnose prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate accuracy of the new image-guided targeted needle biopsy using the ex-vivo human prostate as obtained from fresh radical prostatectomy specimens.

OUTLINE: Patients undergo robotic radical prostatectomy, followed by 3 MRI-TRUS fusion image-guided prostate biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have biopsy-proven prostate cancer, or prostate-specific antigen (PSA) >= 4 ng/ml or an abnormal digital rectal examination (DRE) if consented before prostate biopsy
* Subjects must have at least 2, preferably 3, pre-operative magnetic resonance imaging (MRI)-identified malignant or benign lesions that measure between 10 mm and 15 mm in diameter within the prostate
* Subjects must have decided to have their prostate surgically removed

Exclusion Criteria:

* Patients who do not give informed consent
* Patients with extracapsular extension of their prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of times the first biopsy needle is placed within 3.0 mm of the center lesion | One month after last patient enrolled is taken off study
  A likelihood ratio test will be used to test for independence among lesions within a prostate (corresponding to a lack of systematic MRI-TRUS image distortion and implying that, overall, 1st biopsies to a lesion within one prostate are as likely to accurate as in another prostate).
Number of times the second biopsy needle is placed within 3.0 mm of the center lesion | One month after last patient enrolled is take off study
  A likelihood ratio test will be used to test for independence among lesions within a prostate (corresponding to a lack of systematic MRI-TRUS image distortion and implying that, overall, 1st biopsies to a lesion within one prostate are as likely to accurate as in another prostate).

SECONDARY OUTCOMES:
Average distance of the first needle to the center of the lesion | One month after last patient enrolled is taken off study
  A nested (random effects) analysis of variance (ANOVA) will be used to analyze the distance of the first needle from the center of the lesion. Standard error or 95% confidence interval will be calculated.
Average distance of the second needle from the first needle minus 2.0 mm | One month after last patient enrolled is taken off study
  A nested (random effects) ANOVA will be used to analyze the distance of the first needle from the center of the lesion.
Average distance of the third needle from the first needle minus 2.0 mm | One month after last patient enrolled is taken off study
  A nested (random effects) ANOVA will be used to analyze the distance of the first needle from the center of the lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Ukimura, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States